CLINICAL TRIAL: NCT02904317
Title: The Misoprostol Vaginal Insert Compared With Oral Misoprostol for Labour Induction in Term Pregnancies: a Pair-matched Case-control Study
Brief Title: Misoprostol for Labour Induction
Status: Completed | Type: Observational
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Principal Investigator, Peter Schwaerzler, Principal investigator, Asklepios Kliniken Hamburg GmbH
Other Study IDs: PV4803-2
Record Dates: First submitted 2016-08-03; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Labour Induction

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Misprostol vaginal insert for labour induction: 69 patients matching the inclusion criteria and received MVI for labour induction
- Oral misoprostol for labour induction: 69 patients matching the inclusion criteria and received OM for labour induction

SUMMARY:
Objective: To compare the efficacy and safety of the misoprostol vaginal insert (MVI) with an off-label use of oral misoprostol (OM).

Design: Pair-matched case-control study.

Setting: Tertiary-care academic centre in Germany.

Population: A cohort of 138 women ≥ 37/0 weeks pregnant undergoing labour induction.

Methods: The induction of labour with a retrievable prostaglandin vaginal insert in a consecutive series of 69 women was compared with induction using oral misoprostol in a pair-matched cohort.

Main outcome measures: The primary outcomes were the time from induction to delivery and the caesarean section rate. Secondary outcomes included uterine tachysystole, tocolysis, fetal scalp blood testing, meconium-stained amniotic fluid, umbilical arterial pH, and Apgar score.

DETAILED DESCRIPTION:
Open, non-interventional study in a tertiary referral center in Germany N/A The rationale of our observational study is to describe the efficacy and safety profile of the drug with definition of active labor according to local clinical practice in a descriptive observational study in a tertiary referral center.

A time interval from induction of labor to delivery is depending on the duration of the MISODEL® application. By an observational study the investigators want to describe the efficacy and safety with regard to time to delivery and complication rate.

Primary Objective:

The aim of this study is to describe time to vaginal delivery with definition of active labor according to local clinical practice.

The time period needed to induce any delivery and to describe the drug safety profile.

Primary endpoints:

* Time to vaginal delivery in hours in patients with vaginal delivery.
* Length of time until any delivery
* Caesarean section rate
* Time until onset of labor
* Frequency of vaginal operative delivery
* Frequency of abnormal CTG (Figo)
* Frequency of uterine Tachysystole leading to abnormal fetal heartrate i.e. Figo P. Tachysystole is defined as five or more contractions in 10 minutes averaged over three consecutive 10-minute periods.
* Written informed consent of the patients
* ≥18 years of age
* Parity five or less with singleton pregnancies
* ≥36 weeks of gestation
* Unfavourable cervix (baseline modified Bishop score ≤6)

Misoprostol 200mcg VDS is contraindicated according to the SmPC in the following cases:

* When there is hypersensitivity to the active substance or to any of the excipients
* When labour has started
* When oxytocic drugs and/or other labour induction agents are being given
* When there is suspicion or evidence of uterine scar resulting from previous uterine surgery, e.g. C-section
* When there is uterine abnormality (e.g. bicornate uterus)
* When there is placenta praevia or unexplained vaginal bleeding after 24 weeks gestation with this pregnancy
* When there is foetal malpresentation
* When there are signs or symptoms of chorioamnionitis, unless adequate prior treatment has been instituted
* Before week 36 of gestation

For evaluation of the primary and secondary endpoints of the study, descriptive statistical methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* gynaecologist's indication for induction
* informed consent
* > 37 weeks of gestation
* singleton pregnancies
* cephalic presentation
* cervical Bishop score of < 5 before priming reassuring fetal heart rate

Exclusion Criteria:

* known hypersensitivity to prostaglandins
* uterine scar
* parity > 5
* any contraindication for vaginal delivery
* cephalopelvic disproportion
* placenta previa
* chorioamnionitis
* antepartum bleeding of unknown aetiology
* cardiopulmonary, renal, hepatic maternal disease glaucoma
* fetal congenital abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 138 women ≥ 37/0 weeks pregnant undergoing labour induction.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
time from application of the medication until delivery in minutes | September 2015

SECONDARY OUTCOMES:
Rate of participants receiving a caesarean section compared to all participants being induced | September 2015
Number of participants with treatment-related tachysystole as assessed by cardiotocography | September 2015
Number of participants with treatment-related adverse events following tocolysis with Partusisten | September 2015
Number of participants with fetal compromise assessed by the APGAR-Score and the postpartum fetal pH-value | September 2015

IPD SHARING:
Plan to Share IPD: No